CLINICAL TRIAL: NCT04239781
Title: A Questionnaire Survey for Factors That Influence Postoperative Treatment Decision-making in Patients With Hepatocellular Carcinoma
Brief Title: A Survey for Factors That Influence Postoperative Treatment Decision-making for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Professor of Surgery, Shanghai Zhongshan Hospital
Other Study IDs: HCC treatment survey
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional and questionnaire survey study. The investigators try to find out patient's willingness and expectation for post-operative treatments for hepatocellular carcinoma (HCC), as well as patients' willingness to participate in clinical trials using a questionnaire. The ultimate goal is to assist physicians in clinical treatment decision, clinical research, and government health and economic decision-making, as well as to help investigators understand how to increase public awareness of the HCC and the treatment course and efficacy of HCC, and the awareness of clinical trials.

DETAILED DESCRIPTION:
There is no world widely accepted adjuvant therapy for HCC and the guidelines from AASLD or EASL did not recommend any adjuvant therapy to prevent postoperative tumor recurrence of HCC. The goal of an adjuvant therapy is to meet the requirements of patients, which are influenced by many factors such as the strength of doctors' recommendation, economic affordability, tolerance of adverse reactions to treatment, and expectation of efficacy. Therefore, understanding patients' expectations for an adjuvant therapy after surgery will help doctors give more reasonable treatment. Participating in clinical trials is a new process of understanding and acceptance for each patient, so investigators try to understand the willingness and ideas of patients to participate in clinical trials, so as to provide more information for designing clinical trials and recruiting subjects for clinical trials.

The research was conducted through face-to-face interview, WeChat and telephone interview. For face-to-face interview and WeChat to participants, an informed consent should be signed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older;
* Confirmed diagnosis of HCC histologically or clinically;
* The participant must have received surgical resection;
* Ability to complete the questionnaire or independently or with the help of a friend, relative, or staff member of the oncology department.

Exclusion Criteria:

* The patients that researchers consider not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received surgical resection for hepatocellular carcinoma or their relatives
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
HCC patients' willingness and expectation for post-operative treatment. | 6 months
  Use questionnaires to understand the willingness and expectation of patients for post-operative treatment of hepatocellular carcinoma, as well as their willingness to participate in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Huichuan Sun, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No